CLINICAL TRIAL: NCT06565819
Title: A Trial of Important Parameters of NIR-II Imaging in the Diagnosis of Lower Extremity Peripheral Artery Disease in Patients With Type 2 Diabetes
Brief Title: Important Parameters of NIR-II Imaging in the Early Diagnosis of Lower Extremity Peripheral Artery Disease
Status: Completed | Type: Observational
Sponsor: Yijie Ning (Other)
Responsible Party: Sponsor-Investigator, Yijie Ning, Doctor of vascular surgery, Second Hospital of Shanxi Medical University
Organization: Second Hospital of Shanxi Medical University (Other)
Other Study IDs: [2024]YX211
Record Dates: First submitted 2024-08-14; First posted 2024-08-22 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Peripheral Artery Disease
Keywords: Peripheral artery disease; Second near-infrared region imaging
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Diagnostic Imaging; Ultrasonography, Doppler, Duplex

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with type 2 diabetes who had not been diagnosed with lower peripheral artery disease: Patients received NIR-II and DUS six months and one year after the first NIR-II examination
  Interventions: Diagnostic Test: The second near-infrared region (NIR-II) imaging for lower extremity peripheral artery disease (PAD)

INTERVENTIONS:
Diagnostic Test: The second near-infrared region (NIR-II) imaging for lower extremity peripheral artery disease (PAD) — DUS was used as reference criteria to screen out patients newly diagnosed with PAD during follow-up. In this study, NIR-II imaging results of patients at follow-up and initial examination were collected to obtain a threshold for early diagnosis.
  Other Names: Duplex ultrasound (DUS)

SUMMARY:
Lower extremity peripheral artery disease (PAD) is a growing global health problem. New ways have been explored to diagnose PAD in recent years, such as the second near-infrared region (NIR-II, 900-1,880 nm wavelengths) imaging. In this study, NIR-II imaging was performed on patients with type 2 diabetes without PAD, and time-intensity curves were generated according to the imaging results, and specific parameters on the curves were analyzed. The key parameters for the diagnosis of lower limb artery plaque were obtained by comparing the parameters of patients with and without plaque. Patients will be followed up six months and one year after the first NIR-II imaging. The patient will undergo Duplex ultrasound (DUS), NIR-II imaging and laboratory examination. With DUS results as the reference standard, patients diagnosed with PAD for the first time during follow-up were focused on, and the parameter range of the first NIR-II imaging was statistically analyzed, so as to obtain the diagnostic threshold for early diagnosis of PAD.

DETAILED DESCRIPTION:
1. The registry procedures and quality assurance: the study recruited patients diagnosed with type 2 diabetes from the Department of Endocrinology at the Second Hospital of Shanxi Medical University. If the patient meets the inclusion criteria and agrees to be enrolled, a written informed consent will be signed. The imaging process is completed by a uniform standard, and all imaging operations are performed by the same operator. The operator has been formally trained and the procedure and results are checked by another professional NIR imaging engineer.
2. Imaging process: The imaging device used was Full Spectrum Opening in Vivo Fluorescence Imaging System (DPM-IVFM-NIR-OF, Beijing Digital Precision Medicine Technology Co., Ltd., China). Firstly, participants were asked if they had a history of indocyanine green (ICG) or iodine allergy. If there was no relevant allergy history, an ICG skin test was performed on each participant. The skin test reagent was the ICG solution (Dandong Yichuang Pharmaceutical, China) with a concentration of 0.005mg/mL (diluted with sterile water for injection) . The test reagent (0.1 ml) was injected subcutaneously into the inner forearm and the subject was observed for 20 min. If there was no allergic reaction, an indent needle was placed in the basilic vein of patients. The NIR imaging was conducted in a room without natural light. Before the examination, the subject rested for at least 15 min in a supine position with both knee joints bent 90 degrees and both feet put together, and then step horizontally on the black background board on the examination bed. In NIR-II imaging, the selected filter was 1000 nm long-pass. The power of the 808nm wavelength laser emitter was adjusted to 10000mW with the aperture size adjusted to 2.0 and the exposure time set to 100 ms. The laser emitter was fixed at 20cm vertical to the dorsal foot, and the NIR-II camera was fixed at 40cm vertical to the dorsal foot. ICG solution (2.5 mg/mL, diluted with sterile water for injection) was administered intravenously via an indignant needle. The dose of ICG injected was determined according to body weight: 0.1mg/Kg. The time for intravenous injection of ICG solution was 5 seconds. The intensity of fluorescence signal on both the dorsal feet was recorded within 5 minutes after ICG solution was injected. The dorsal pedis region from the transverse tarsus joint to the distal metatarsal bone was selected as the region of interest (ROI). The ROI was analyzed using the built-in analysis software External Data processing to generate a time-intensity curve.
3. Plan for missing data: missing data will be excluded from analysis.
4. Methods to summarize the data: NIR-II parameters extracted from time-intensity curves for all patients were recorded in the same excell table. In addition, baseline information (such as age, gender, height, weight, etc.) and clinical characteristics (such as years of diabetes, hypertension, hyperlipidemia, etc.) of all patients were recorded in this table.
5. Statistical analysis: In this study, SPSS 26.0 software and R 4.2.0 software were used to conduct in-depth statistical research. When processing measurement data, the Kolmogorov-Smirnov test was first used to verify whether the data followed the normal distribution. Data with a normal distribution was represented by x±s, while data with a skewed distribution was represented by M (Q1, Q3). For comparison between groups, the independent sample test or the Mann-Whitney U test were selected. For classified data, χ2 test or Fisher exact probability method was chosen for further investigation. A significance level of P < 0.05 means that the difference was statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects are inpatients in the Department of Endocrinology, the Second Hospital of Shanxi Medical University.
2. Male or female aged 18-85.
3. Patients with type 2 diabetes (WHO 2019 diagnostic criteria).
4. The subjects are conscious and fully aware of the research content. They sign the informed consent and agree to participate in the study.

Exclusion Criteria:

1. The patients who have been diagnosed with thyroid disease or are using other drugs that affect metabolism and cannot stop taking them.
2. Indocyanine green or iodine allergy
3. Previous history of lower limb revascularization surgery or lower limb amputation, or diabetic foot ulcers (current or past).
4. Lymphedema, thrombophlebitis, deep vein thrombosis (current or past 6 months).
5. Patients with acute infections, tumors, severe arrhythmias, psychiatric disorders, drug or alcohol addiction.
6. NYHA grade Ⅱ - Ⅳ heart failure, liver function significantly abnormal or kidney function significantly abnormal
7. Pregnant women, women planning pregnancy or breastfeeding.
8. Participated in other clinical trials within 3 months prior to the trial.
9. Refuse to sign informed consent and agree to participate in this study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population were inpatients with type 2 diabetes from the Department of Endocrinology, the Second Hospital of Shanxi Medical University.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2024-09-15 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Time related NIR-II parameters for patients newly diagnosed with PAD during follow-up (parameters at first imaging and follow-up imaging) | Baseline, 6 months and 1year
  In this study, 5-minute NIR-II imaging video of each patient was processed into time-intensity curves to quantify the imaging results. Four time related parameters on time-intensity curves were extracted, including：T start (s), Tmax (s), T 1/2 (s), TR (Time ratio).
  Note: "s" is used as the unit "second".
Intensity related NIR-II parameters for patients newly diagnosed with PAD during follow-up (parameters at first imaging and follow-up imaging) | Baseline, 6 months and 1year
  In this study, 5-minute NIR-II imaging video of each patient was processed into time-intensity curves to quantify the imaging results. Three intensity related parameters on time-intensity curves were extracted, including：Imax (Fi), Ingress (Fi), Engress (Fi).
  Note: "Fi" is used as the unit "fluorescence intensity".
Time-intensity related NIR-II parameters for patients newly diagnosed with PAD during follow-up (parameters at first imaging and follow-up imaging) | Baseline, 6 months and 1year
  In this study, 5-minute NIR-II imaging video of each patient was processed into time-intensity curves to quantify the imaging results. Two time-intensity related parameters on time-intensity curves were extracted, including：Ingress rate (Fi/s), Engress rate (Fi/s).
  Note: "s" is used as the unit "second" and "Fi" is used as the unit "fluorescence intensity".

CONTACTS AND LOCATIONS:
Overall Officials: Ruijing Zhang, Doctoral degree, Study Director — Second Hospital of Shanxi Medical University; Honglin Dong, Doctoral degree, Study Chair — Second Hospital of Shanxi Medical University
Locations (1):
- Full Spectrum Opening in Vivo Fluorescence Imaging System (DPM-IVFM-NIR-OF, Beijing Digital Precision Medicine Technology Co., Ltd., China), Taiyuan, Shanxi, China

IPD SHARING:
Plan to Share IPD: Yes
Patient baseline data and statistical methods will be shared
Supporting Information: SAP
Time Frame: Starting 1 year after publication
Access Criteria: If there are researchers who need to get the shared data, please contact Yijie Ning via email and explain the purpose of using the data. We will send the shared data to your email.

REFERENCES:
- [Result] van den Hoven P, Ooms S, van Manen L, van der Bogt KEA, van Schaik J, Hamming JF, Vahrmeijer AL, van der Vorst JR, Mieog JSD. A systematic review of the use of near-infrared fluorescence imaging in patients with peripheral artery disease. J Vasc Surg. 2019 Jul;70(1):286-297.e1. doi: 10.1016/j.jvs.2018.11.023. PMID 31230648
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/31230648/